CLINICAL TRIAL: NCT03421509
Title: The Association Between Cutaneous Silent Period Parameters and Spasticity in Patients With Stroke
Brief Title: Cutaneous Silent Period and Spasticity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2017.679
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Stroke
Keywords: cutaneous silent period; spasticity; stroke
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cutaneous silent period — In the upper limb the cutaneous silent period (CSP) is a brief transient suppression of the voluntary muscle contraction that follows painful stimulation applied to the finger (digits II-V, C6-C8 dermatomes)

SUMMARY:
The cutaneous silent period (CSP) is a brief transient suppression of the voluntary muscle contraction that follows a noxious cutaneous nerve stimulation. Studies in patients with central disorders of motor control such as dystonia and Parkinson's disease have shown CSP abnormalities indicating that supraspinal pathways influence this inhibitory spinal reflex. The aim of this study is to investigate the association between CSP parameters (duration and latency) and spasticity in stroke.

DETAILED DESCRIPTION:
The cutaneous silent period (CSP) is a brief transient suppression of the voluntary muscle contraction that follows a noxious cutaneous nerve stimulation. Studies in patients with central disorders of motor control such as dystonia and Parkinson's disease have shown CSP abnormalities indicating that supraspinal pathways influence this inhibitory spinal reflex. Spasticity is a serious problem that creates great difficulty for both patients and clinicians. The Support Programme for Assembly of a database for Spasticity Measurement (SPASM) group defined the spasticity as "disordered sensory-motor control, resulting from an upper motor neuron lesion, presenting as intermittent or sustained involuntary activation of muscles". Spasticity occurs in different types depending on the duration of the lesion present in the central nervous system (acute or slowly emerging), the size of the lesion and the location of the lesion such as cerebral cortex, brain stem or spinal cord. There are three major approaches, clinical, neurophysiological and biomechanical, for assessing spasticity. Stimulating the cutaneous nerve of the index finger at low-intensity, researchers have evoked an inhibition of the electromyographic (EMG) activity with a long latency and a short duration, namely the I2 inhibitory response of the cutaneo-muscular reflexes in the hand. ıt was suggested that the I2 inhibitory response, whose latency and duration overlap the CSP, was mediated by low-threshold, large-diameter fibers. Hence, because high-intensity electrical stimuli used to evoke the CSP activate large-diameter as well as small-diameter fibers, both fiber types may contribute in generating the CSP .

The central neural substrates producing the alpha-motor neuron inhibition after high-intensity stimulation differ from those after low-intensity stimulation. Low-intensity non-painful stimulation elicits a typical polysynaptic pattern of exteroceptive reflexes, whereas high-intensity electrical stimulation elicits an oligosynaptic pattern. Several studies investigated whether the CSP after high intensity finger stimulation arises from interruption of the excitatory drive to motor neurons (pre-synaptic inhibition) or inhibition of motor neurons themselves (post-synaptic inhibition). Studies using H-reflexes, F waves, and motor evoked potentials to assess motor neuron excitability showed that during the CSP motor neurons mainly receive post-synaptic inhibition transmitted through spinal inhibitory interneurons. Studies in patients with central disorders of motor control such as dystonia and Parkinson's disease have shown CSP abnormalities indicating that supraspinal pathways influence this inhibitory spinal reflex.

It was investigated whether the CSP parameters, F parameters are different between patients with stroke and amyotrophic lateral sclerosis (ALS) and healthy controls.

They found that CSP latency was higher in patients with stroke and ALS than healthy subjects. There was no difference in KSP duration and F-latency compared to healthy subjects. Contrary to these results, in another study did not show a relationship between spasticity and CSP parameters in twelve patients with stroke. The results of the existing studies on the relationship between spasticity and CSP parameters are conflicting. The influence of the descending suprasegmental pathways on the origin of the CSP is yet to be elucidated. Therefore; there is a need for a properly designed study investigating this relationship in a homogeneous sample. Given these results, we aimed to investigate the association between CSP parameters (duration and latency) and spasticity in patients with stroke. modified Ashworth scale, Modified Tardieu scale, Brunnstrom motor stage ve Fugl Meyer upper extremity score, Barthel index will be measured. Patients with stroke will underwent electromyographic assessments of F-wave latency, F-M ratio, CSP latency and duration, upper extremity nerve conduction studies. Association between clinical assessments and electrophysiological assessments will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. First ever time stroke
2. Time since stroke >1 month
3. Being able to understand the instructions (mini mental test score>24)

Exclusion Criteria:

1. Diseases which might affect CSP parameters (Parkinsonism, restless leg syndrome, carpal tunel syndrome etc.)
2. Autonomic nervous system disease
3. Antispasticity medication use
4. Hemiplegic shoulder pain
5. Botulinum toxin injection within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-70 years old patients with stroke will be allowed.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Cutaneous silent period latency (ms) | Day 1
  the brief interruption in voluntary contraction that follows strong electrical stimulation (painful) of a cutaneous nerve. time between the stimulation and beginning of the silent period.
Cutaneous silent period duration (ms) | Day 1
  the brief interruption in voluntary contraction that follows strong electrical stimulation (painful) of a cutaneous nerve. CSP duration is defined as the time between the beginning and endpoint of the silent period

SECONDARY OUTCOMES:
Modified Ashworth Scale wrist | Day 1
  Scores range from 0-4, with 5 choices 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement) 2 (3) - More marked increase in musce tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale finger flexors | Day 1
  Scores range from 0-4, with 5 choices 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement) 2 (3) - More marked increase in musce tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Tardieu Scale R1 wrist | Day 1
  The angle of full ROM (R2) is taken at a very slow speed (V1). The angle of muscle reaction (R1) is defined as the angle in which a catch or clonus is found during a quick stretch (V3). R1 is then subtracted from R2 and this represents the dynamic tone component of the muscle
Modified Tardieu Scale R1 finger flexors | Day 1
  The angle of full ROM (R2) is taken at a very slow speed (V1). The angle of muscle reaction (R1) is defined as the angle in which a catch or clonus is found during a quick stretch (V3). R1 is then subtracted from R2 and this represents the dynamic tone component of the muscle
Modified Tardieu Scale R2 wrist | Day 1
  The angle of full ROM (R2) is taken at a very slow speed (V1). The angle of muscle reaction (R1) is defined as the angle in which a catch or clonus is found during a quick stretch (V3). R1 is then subtracted from R2 and this represents the dynamic tone component of the muscle
Modified Tardieu Scale R2 finger flexors | Day 1
  The angle of full ROM (R2) is taken at a very slow speed (V1). The angle of muscle reaction (R1) is defined as the angle in which a catch or clonus is found during a quick stretch (V3). R1 is then subtracted from R2 and this represents the dynamic tone component of the muscle
Modified Tardieu Scale R2-R1 wrist | Day 1
  The angle of full ROM (R2) is taken at a very slow speed (V1). The angle of muscle reaction (R1) is defined as the angle in which a catch or clonus is found during a quick stretch (V3). R1 is then subtracted from R2 and this represents the dynamic tone component of the muscle
Modified Tardieu Scale R2-R1 finger flexors | Day 1
  The angle of full ROM (R2) is taken at a very slow speed (V1). The angle of muscle reaction (R1) is defined as the angle in which a catch or clonus is found during a quick stretch (V3). R1 is then subtracted from R2 and this represents the dynamic tone component of the muscle
Brunnstrom stage arm | Day 1
  Motor recovery stage after stroke The Seven Brunnstrom Stages of Motor Recovery (see table below for more details)
  1. Flaccid paralysis. No reflexes.
  2. Some spastic tone. No voluntary movement. Synergies elicited through facilitation.
  3. Spasticity is marked. Synergistic movements may be elicited voluntarily.
  4. Spasticity decreases. Synergistic movements predominate.
  5. Spasticity wanes. Can move out of synergies although synergies still present.
  6. Coordination and movement patterns near normal. Trouble with more rapid complex movements.
  7. Normal.
Brunnstrom stage hand | Day 1
  Motor recovery stage after stroke The Seven Brunnstrom Stages of Motor Recovery (see table below for more details)
  1. Flaccid paralysis. No reflexes.
  2. Some spastic tone. No voluntary movement. Synergies elicited through facilitation.
  3. Spasticity is marked. Synergistic movements may be elicited voluntarily.
  4. Spasticity decreases. Synergistic movements predominate.
  5. Spasticity wanes. Can move out of synergies although synergies still present.
  6. Coordination and movement patterns near normal. Trouble with more rapid complex movements.
  7. Normal.
Fugl Meyer upper extremity score | Day 1
  Items are scored on a 3-point ordinal scale 0 = cannot perform
  1. = performs partially
  2. = performs fully Maximum score=66
Barthel index | Day 1
  ordinal scale used to measure performance in activities of daily living (ADL) Minimum-maximum score: 0-100
F wave latency | Day 1
  the time from the onset of the stimulation artifact to the first deflection of the waveform from baseline <32 ms when obtained from median/ulnar nerves
F/M ratio | Day 1
  The F/M ratio compares proximal and distal segments and is useful in evaluating conduction time from stimulation site to spinal cord

CONTACTS AND LOCATIONS:
Overall Officials: Gulseren Derya AKYÜZ, Prof, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Floeter MK. Cutaneous silent periods. Muscle Nerve. 2003 Oct;28(4):391-401. doi: 10.1002/mus.10447. PMID 14506711
- [Background] Gilio F, Bettolo CM, Conte A, Iacovelli E, Frasca V, Serrao M, Giacomelli E, Gabriele M, Prencipe M, Inghilleri M. Influence of the corticospinal tract on the cutaneous silent period: a study in patients with pyramidal syndrome. Neurosci Lett. 2008 Mar 12;433(2):109-13. doi: 10.1016/j.neulet.2007.12.055. Epub 2008 Jan 10. PMID 18242857
- [Background] Kwang-Ik Jung WK. The Relationship between Cutaneous Silent Period and Spasticity in Patients with Stroke. Jouranl of Korean Association of EMG Electrodiagnostic Medicine, 10( 1), 1- 5. 2008.
- [Background] Naghdi S, Ansari NN, Abolhasani H, Mansouri K, Ghotbi N, Hasson S. Electrophysiological evaluation of the Modified Tardieu Scale (MTS) in assessing poststroke wrist flexor spasticity. NeuroRehabilitation. 2014;34(1):177-84. doi: 10.3233/NRE-131016. PMID 24284462